CLINICAL TRIAL: NCT03831269
Title: Role of Streptococcal Infection in the Etiopathogenesis of Pityriasis Lichenoides Chronica and the Therapeutic Efficacy of Azithromycin; a Randomized Controlled Trial
Brief Title: Pityriasis Lichenoides Chronica, Role of Streptococcal Infection and Azithromycin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Elbendary, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kasr Alainy Cairo U
Record Dates: First submitted 2019-01-25; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Pityriasis Lichenoides
MeSH Terms: conditions — Pityriasis Lichenoides | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin (Active Comparator): The dose of azithromycin will be 10mg/kg/day oral suspension for 3 consecutive days for pediatric patients (<12 years old) and 500mg/day in three consecutive days for adults. The cycle will be repeated every seven days (3 cycles/month) and will be repeated if required according to patient's response up to 6 cycles. Side effects of therapy will be recorded. This protocol is based on previous case reports.
  Interventions: Drug: Azithromycin
- Nb UVB (Active Comparator): Patients recruited for nbUVB phototherapy will have an initial dose of 0.3J-0.5J according to Fitzpatrick's skin type. The dosage will be increased by 0.3J in every other treatment session. The sessions will be given 3 times weekly until improvement is noted or reaching 8 weeks at the EOS. We arrived at this initial dose based on our previous experience with Egyptian patients in Kasr Alainy phototherapy unit in Dermatology Department, Cairo University.
  Interventions: Other: nbUVB

INTERVENTIONS:
Drug: Azithromycin — Patients will be randomly distributed and start taking azithromycin according to the known dose /kg/day for repeated cycles till improvement or reaching the end of study
  Arms: Azithromycin
Other: nbUVB — The patients will be randomly distributed to start nbUVB sessions and clinical improvement will be compared to that of Azithromycin
  Arms: Nb UVB

SUMMARY:
Primary outcome:

The primary outcome at end of study (EOS) is to compare the therapeutic efficacy of Azithromycin in the treatment of pityriasis lichenoides chronica (PLC) with that of a well-documented line of therapy namely narrow band ultra violet B (nbUVB).

Secondary outcomes:

1. To identify the possibility of streptococcal throat infection as a possible underlying etiology in PLC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with classic papular eruption of PLC (scaly erythematous papules with mica-like scales) with diagnosis documented histopathologically with or without associated hypopigmented lesions
2. Age: > 6 years
3. Both sexes.

Exclusion Criteria:

1. Patients presenting with only hypopigmented macules whom their skin biopsy revealed PLC.
2. Patients with hypopigmented lesions that reveal mycosis fungoides pathologically.
3. Patients with PLC associated with classic MF.
4. Patients with known absolute contraindications to NB-UVB.
5. Patients with impaired liver and/or kidney functions.
6. Patients with history of any heart disease.
7. Patients with known hypersensitivity to Azithromycin

   -

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Azithromycin in treating pityriasis lichenoides chronica | 12 months
  The clinical improvement of patients with PLC will be evaluated after taking 3 to 6 cycles of azithromycin and will be compared to the clinical outcome of patients that had three sessions of nbUVB for six to eight weeks. Side effects will be documented in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Faculty of Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Email contact

REFERENCES:
- [Derived] Elbendary A, Youssef R, Abdel-Halim MRE, Abdel Halim D, El Sharkawy DA, Alfishawy M, Gad MA, Gad A, Elmasry MF. Role of streptococcal infection in the etiopathogenesis of pityriasis lichenoides chronica and the therapeutic efficacy of azithromycin: a randomized controlled trial. Arch Dermatol Res. 2023 Apr;315(3):521-530. doi: 10.1007/s00403-022-02398-0. Epub 2022 Sep 21. PMID 36129521